CLINICAL TRIAL: NCT05736575
Title: Differences in Brain Derived Neurotrophic Factor Levels Between Chronic and Asymptomatic Pain Patients
Acronym: BDNF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal Investigator, Universidad Autonoma de Madrid
Other Study IDs: CCBDNF
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain
Keywords: BDNF
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — BDNF levels will be measured through a blood sample taken by a nurse and analysed by a biochemist. Blood collection has been chosen over saliva analysis because the former has been shown to be the most reliable method for measuring this neurotrophin at the peripheral level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Pain Patient: A blood draw is to be performed to analyze peripheral BDNF.
  Interventions: Genetic: BDNF analysis (Elisa KIT)
- Asymptomatic subject: A blood draw is to be performed to analyze peripheral BDNF.
  Interventions: Genetic: BDNF analysis (Elisa KIT)

INTERVENTIONS:
Genetic: BDNF analysis (Elisa KIT) — Analysis of peripheral BDNF will be performed

SUMMARY:
A case-control study will be conducted to analyze the differences in BDNF levels between patients with chronic pain and asymptomatic people.

DETAILED DESCRIPTION:
Brain-derived neurotrophic factor (BDNF) is considered a biomarker of brain plasticity. Since different alterations in brain plasticity have been found in chronic pain patients, the investigators want to study whether there are differences at the molecular level in this population compared to an asymptomatic population in order to be able to accurately measure the impact of different physiotherapy interventions in an objective way.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18 to 65 years with musculoskeletal pain for a minimum of 3 months
* patients recruited by information pamphlets from the university clinic of the Rey Juan Carlos University, and CSEU La Salle
* not having received physiotherapy treatment for this same process in the last 3 months.
* ability to perform all the clinical tests and to understand the study process, as well as to obtain informed consent.

Exclusion Criteria:

* Systemic, neurological, oncological or inflammatory diseases; psychiatric pathologies, pregnancy, type II diabetes.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: subjects will be selected if they have been suffering from musculoskeletal pain (not oncological) for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
BDNF Levels | 3 hours
  Brain Derived Neurotrophic Factor: Pierce NeutrAvidin-coated high-capacity plates (ThermoFisher Scientific; 15509) will incubate for two hours at RT with 200 µl of 14 µg/ml biotin-conjugated mAb-#1 diluted in phosphate buffer (0.1% Triton X-100 in 0.1 M phosphate buffer: 0.1 M KH2PO4 and 0.1 M Na2HPO4; pH 7.6). Plates will then washed three times with blocking buffer [1% bovine serum albumin (BSA); Sigma A2153 in phosphate buffer], followed by the addition of 150 µl phosphate buffer. A total of 50 µl of either standards or diluted samples (both in blocking buffer) will then added to the plate followed by incubation for 3 h at RT on a rotary shaker.
Pain Intensity | 3 hours
  Pain intensity assessed with the 100 mm Visual Analog Scale, in which the patient is asked about his or her pain level at that moment, with one side being "no pain" and the other extreme being "the worst pain imaginable"

CONTACTS AND LOCATIONS:
Locations (1):
- Irf Cseuls, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No